CLINICAL TRIAL: NCT01750216
Title: An Observational Study of Peginterferon-alfa-2a (Pegasys) and Ribavirin (Copegus) on Predictive Values of RVR on Sustained Virological Response (SVR) in Different Stage of Liver Fibrosis in Treatment-naïve Patients With Genotype 1 Chronic Hepatitis C
Brief Title: An Observational Study of Pegasys (Peginterferon Alfa-2a) and Copegus (Ribavirin) on Predictive Values of RVR on Sustained Virological Response in Different Stages of Liver Fibrosis in Treatment-Naïve Patients With Chronic Hepatitis C Genotype 1
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28344
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the predictive value of rapid virological response (RVR) and early virological response (EVR) on sustained virological response (SVR) by stage of liver fibrosis in treatment-naïve patients with chronic hepatitis C genotype 1 initiated on treatment with Pegasys (peginterferon alfa-2a) and Copegus (ribavirin). Patients will be followed for 48 weeks of treatment and up to 24 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Chronic hepatitis C genotype 1
* Treatment-naïve, i.e. have not been previously treated with pegylated interferon, standard interferon and ribavirin
* Confirmed serum positive HCV RNA
* Liver fibrosis confirmed histologically or by fibroscan up to 24 months before treatment

Exclusion Criteria:

* Any contraindications according to the Summary of Product Characteristics for Pegasys or Copegus
* Co-infection with hepatitis B or HIV
* Post-transplant patients
* End stage renal disease (creatinine clearance < 15 ml/min)
* Patients treated with immunotherapy
* Pregnant women and male partners of women who are pregnant
* Female patients of childbearing potential and male patients with female partners of childbearing potential who are unable or unwilling to use effective and continuous contraception during the treatment and for 4 months (females) and 7 months (males) thereafter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve patients with chronic hepatitis C genotype 1 initiated on treatment with Pegasys and Copegus
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Sustained virological response (SVR) rate, in relation to rapid virological response (RVR) in different stages of liver fibrosis in treatment-naïve patients with chronic hepatitis C genotype 1 | approximately 3 years

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | approximately 3 years
Sustained virological response (SVR) rate, in relation to early virological response (EVR) in different stages of liver fibrosis in treatment naïve patients with chronic hepatitis C genotype 1 | approximately 3 years
Response rates (RVR, EVR, SVR) according to host/virus/treatment-related factors in different stages of liver fibrosis (F>/=3 and </=3) | approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Poland (14):
  - Bydgoszcz
  - Bytom
  - Chorzów
  - Ciechanów
  - Dębica
  - Katowice
  - Koszalin
  - Lodz
  - Mielec
  - Puławy
  - Radom
  - Warsaw
  - Wałbrzych
  - Łańcut